CLINICAL TRIAL: NCT06584149
Title: The Role of Blood Urea Nitrogen to Serum Albumin Ratio in the Prediction of Mortality in Septic Acute Kidney Injury Patients
Brief Title: BAR As a Mortality Predictor in Septic AKI
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: BAR in septic AKI
Record Dates: First submitted 2024-08-24; First posted 2024-09-04 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury; Sepsis
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to investigate the prognostic value of Blood Urea Nitrogen to serum Albumin ratio in septic Acute Kidney Injury patients Follow-up will be conducted for all enrolled patients for 30 days from admission to record mortality and the cause of death.

DETAILED DESCRIPTION:
A complete medical history will be obtained from all patients including age, sex, comorbidities, cause of sepsis, and SOFA and APACHE II scores at admission.

Blood samples will be collected within 24 hours of AKI diagnosis for analysis of Blood Urea Nitrogen (BUN) and serum Albumin levels.

Blood Urea Nitrogen to serum Albumin ratio (B/A) will be calculated by dividing the BUN of a patient by their serum Albumin levels.

Laboratory parameters also will include pH, lactate (Lac), base excess (BE), hemoglobin (Hb), platelet (PLT) count, white blood cell (WBC) count, bilirubin, hematocrit (HCT), creatinine (Cr), serum sodium (Na), serum potassium (K), serum calcium (Ca), serum magnesium (Mg), triglyceride (TG), aspartate aminotransferase (ALT), alanine aminotransferase (AST), prothrombin time (PT), and activated partial thromboplastin time (APTT) values.

Follow-up will be conducted for all enrolled patients for 30 days from admission to record mortality and the cause of death.

Study population will be divided into survival and non-survival groups based on their 30-day survival status

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 60 years of age
2. Fulfilled the diagnostic criteria of Sepsis 3.0 (defined as a suspected or confirmed infection with a sequential organ failure assessment (SOFA) score of 2 or higher)
3. Developed AKI during hospitalization according to Kidney Disease: Improving Global Outcomes (KDIGO) guideline

Exclusion Criteria:

1. ICU length of stay<24 h
2. AKI occurred before current hospital admission.
3. AKI is supposed to be secondary to causes other than sepsis.
4. Receiving renal replacement therapy at the time of admission.
5. Diagnosis with chronic kidney disease.
6. Diagnosis with liver failure.
7. Pregnant or lactating.
8. There was insufficient data for analysis.
9. Patients who had received Human serum Albumin infusion 3 days before ICU admission.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This prospective study will be conducted on patients with septic acute kidney injury. After admission of the patient to ICU in Ain Shams University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
mortality | 30 days
  number of cases of mortality

SECONDARY OUTCOMES:
mechanical ventilation | 30 days
  number of participants who needed mechanical ventilation
stage-3 AKI | 30 days
  number of participants who developed stage-3 AKI
renal replacement therapy | 30 days
  number of participants who needed renal replacement therapy
septic shock | 30 days
  number of participants who developed septic shock
length of ICU stay | 30 days
  length of ICU stay in days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No